CLINICAL TRIAL: NCT00680316
Title: A Phase IV, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Pulmozyme® in 3- to 5-Year-Old Patients With Cystic Fibrosis
Brief Title: A Study of Pulmozyme® (Dornase Alpha) in 3- to 5-Year-Old Patients With Cystic Fibrosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Most patients were unable to perform the test being used to measure lung function, thus it became clear the study would not yield clinically meaningful data
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z4240g
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: Pulmozyme; CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dornase alfa (Experimental)
  Interventions: Drug: Dornase alfa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dornase alfa — 2.5 mL (2.5 mg) dornase alfa nebulized once daily for 16 (+/-2) days
  Other Names: Pulmozyme
  Arms: Dornase alfa
Drug: Placebo — 2.5 mL (2.5 mg) placebo nebulized once daily for 16 (+/-2) days
  Arms: Placebo

SUMMARY:
This was a Phase IV, multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the effect of Pulmozyme on pulmonary function, health-related quality of life (HRQOL), and respiratory symptoms in 3- to 5-year-old children with cystic fibrosis (CF). Approximately 40 patients were planned to be enrolled in this study. However, only 3 patients were eligible for random allocation and received treatment: 1 patient in the Pulmozyme group and 2 patients in the placebo group. All 3 patients completed the study assessments but did not have usable pulmonary function test (PFT) data.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Aged 3-5 years
* Diagnosis of cystic fibrosis

Exclusion Criteria:

* Children taking scheduled inhaled Pulmozyme or hypertonic saline within 56 days prior to Visit 1 or any Pulmozyme in the 28 days before Visit 1
* Involvement in a clinical intervention trial within the 4 weeks prior to Visit 1
* Use of an investigational drug or device within 28 days prior to Visit 1
* Any other condition that might increase the risk of participation to the patient in the judgement of the investigator

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Freemer, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dornase Alfa | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dornase Alfa | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 | 4.6 (1.5) | 4.9 (1.2)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactance at 8 Hz (Xrs8) From Visit 2 to Visit 3 (Change From Baseline at Visit 2 to Visit 3, After Study Drug Treatment).
Description: The fundamental principle of forced oscillometry is that lung function can be assessed by measuring changes in pressure and flow in response to external pressure applied at the airway opening. Reactance is complex measure that incorporates the changes in pressure and volume and the rate of these changes in response to pressure oscillations at a specific frequency. (8Hz was used for the primary endpoint). Reactance is thought to reflect the elastic properties of the lung.
Time Frame: from Visit 2 to Visit 3 (16 +/- 2 days)
Population: Children were unable to perform forced oscillometry (FOT) or did not remain stable during the study. No efficacy analyses were performed because no patients had complete (pre- or post-treatment) data for pulmonary function tests, including FOT.
Arm/Group | Dornase Alfa | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Reactance at 4, 6, and 10 Hz (Xrs4, Xrs6, and Xrs10)
Description: as for outcome 1
Time Frame: from Visit 2 to Visit 3 (16 +/- 2 days)
Population: as for outcome 1
Arm/Group | Dornase Alfa | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Resistance at 4, 6, 8, and 10 Hz (Rrs4, Rrs6, Rrs8, and Rrs10)
Description: The fundamental principle of forced oscillometry is that lung function can be assessed by measuring changes in pressure and flow in response to external pressure applied at the airway opening. Resistance is complex measure that incorporates the lack of changes in pressure and volume and the rate of these changes in response to pressure oscillations at a specific frequency. (10Hz was used for the secondary endpoint).
Time Frame: from Visit 2 to Visit 3 (16 +/- 2 days)
Population: as for outcome 1
Arm/Group | Dornase Alfa | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Respiratory Symptom Domain Score From the Cystic Fibrosis Questionnaire Revised (CFQ-R) for Parents of Preschoolers and for Preschoolers
Description: The CFQ-R for Preschoolers and the CFQ-R for Parents of Preschoolers was designed specifically to measure the impact of CF for patients with a diagnosis of CF. Each question is answered using a 4-point Likert scale.
  In order to calculate the domain/symptom scale scores, the following algorithm is followed
  * Re-number items which have been reverse coded
  * Calculate the mean of the items to be included. If more than half of the items are missing, then the score is considered missing
  * Re-scale to result in a scaled score which ranges from 0 to 100, with higher scores indicating better health
Time Frame: from Visit 2 to Visit 3 (16 +/- 2 days)
Population: as for outcome 1
Arm/Group | Dornase Alfa | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dornase Alfa | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dornase Alfa (N=1) | Placebo (N=2)
Increase in cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bad dreams (Psychiatric disorders) | 0 | 1
Flu symptoms (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Children were unable to perform forced oscillometry (FOT) or did not remain stable during the study. No efficacy analyses were performed because no patients had complete (pre- or post-treatment) data for pulmonary function tests, including FOT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.